CLINICAL TRIAL: NCT00082030
Title: Neural Correlates of Depressive Symptoms and Reward Related Mechanisms Following AMPT Depletion in Remitted Depressed Patients Off Treatment and Healthy Controls
Brief Title: Function of Catecholamines in the Brain During Depression
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040160; 04-M-0160
Record Dates: First submitted 2004-04-28; First posted 2004-04-28 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-11-18

CONDITIONS: Depression; Involutional
Keywords: Depression; PET; fMRI; Dopamine; Norepinephrine Depletion; Emotional Stimuli; Anhedonia; Norepinephrine; Dopamine Depletion; Major Depressive Disorder; MDD; Healthy Volunteer; HV
MeSH Terms: conditions — Depression; Anhedonia; Depressive Disorder, Major

SUMMARY:
This study will explore brain function related to depressive symptoms and will examine DNA for genes that may be involved in depressive disorders, particularly genes that regulate synthesis and metabolism of the brain neurotransmitter catecholamine. It will compare findings in patients with major depressive disorders who are in remission with those in normal, healthy volunteers.

Patients with remitted major depressive disorders and healthy normal volunteers between 18 and 60 years of age may be eligible for this study. Candidates are screened with a psychiatric and medical history, physical examination, electrocardiogram, and blood and urine tests. Participants undergo the following tests and procedures in up to eight visits to the NIH Clinical Center:

Memory Tasks and Problem Solving and Brain Imaging

Subjects are tested with measurements of intelligence or memory ability. They also undergo magnetic resonance imaging (MRI), a test that uses a magnetic field and radio waves to produce images of the brain. For this procedure, the patient lies on a table that is moved into the scanner (a narrow cylinder), and wears earplugs to muffle loud knocking and thumping sounds that occur during the scanning process. The MRI lasts about 60 minutes.

Catecholamine Depletion Study

For this study, subjects take capsules containing either AMPT (a drug that temporarily reduces brain catecholamine activity) or a placebo (lactose capsules, which do not affect brain catecholamine activity) at 9 a.m., 2 p.m., and 7 p.m. on one visit and return the next day to take additional capsules at 7 a.m. and noon. In addition to the study medication, subjects keep a low-monoamine diet (e.g., no chocolate, cheese, smoked meats, and various other foods that will be enumerated) and do not smoke, drink alcohol, or take in food or drink containing caffeine. After taking all the study capsules, the subjects have positron emission tomography (PET) and functional MRI (fMRI) scans, as follows:

* fMRI: While lying in the MRI scanner, the subject performs a monetary reward task that is somewhat like playing a computer video game for money. The amount of cash the subject can win depends on his or her performance. It is possible to lose money that was previously won, if performance declines. This portion of the study provides information on how the brain processes reward and about the role of catecholamines in this process.
* PET: The subject is injected in the arm with a glucose solution that has a radioactive substance attached that can be detected by the PET scanner. During the scan, the subject looks at photographs of faces on a computer screen and is asked to tell the gender of the persons. This test shows brain blood flow and measures brain glucose (sugar) metabolism, which reflects brain activity. At the end of the scan, subjects are asked about their mood and general well being. They return to the Clinical Center the following day for and evaluation of their emotional state.

The catecholamine depletion study is repeated a second time 14 days or more after the first. Subjects who received AMPT capsules for the first study take lactose capsules for the second study, and vice-versa.

DETAILED DESCRIPTION:
The depressive and anhedonic response precipitated by CD raises the possibility that dysfunction of the dopamine system is a stable, sometimes latent characteristic of MDD. Following this line of reasoning, central catecholamine dysfunction as evinced by CD may be equally salient in a subset of unaffected relatives who are at genetic risk for developing the disorder.

We plan to extend the phase I project to unaffected relatives of BD and MDD patients in order to evaluate sensitivity to CD as an endophenotype of MDD and BD. In order to maximize our statistical power, we will be recruiting equal numbers healthy low and high-risk relatives. Here, risk is defined on the basis of chronological age (see below for more detail).

Furthermore, it has recently become feasible to conduct genome-wide association studies and quantify the burden of risk alleles carried by an individual. Certainly, the identity of these risk alleles remains unknown or unproven. Nevertheless, Francis McMahon's group, with whom we are collaborating, have identified upwards of 20 common risk variants in two independent samples. Individuals carrying 19 or more of these risk alleles were found to be 4 times more likely to be cases than controls. This approach may provide us with another method of quantifying genetic risk.

The endophenotypic status of sensitivity to CD will be evaluated with psychometric instruments, FDG PET, and an fMRI-coupled appetitive learning task. We now have access to a high resolution PET scanner (High Resolution Research Tomograph) that will enable us to study hitherto irresolvable structures of importance such as the habenula and peri-aqueductal gray matter (PAG) in addition to previously implicated regions such as the ventral striatum and OFC. Analysis of the metabolic activity of these regions under sham and CD conditions in both remitted MDD and relatives of BD and MDD patients is of great theoretical import. So to is identifying regions of the brain involved in reward response that are selectively impacted by CD, a question that we hope to answer through the use of the fMRI-coupled appetitive learning task.

ELIGIBILITY:
* INCLUSION CRITERIA:

MDD Sample: 40 subjects (ages 18-45) with remitted MDD will be selected. MDD is defined by the DSM-IV criteria, and one of the following additional criteria:

1. history of two or more major depressive episodes, or
2. history of one major depressive episode and a family history for major depression. Remission is defined as a period of at least three months during which the subject has not taken any antidepressant agents, with the Hamilton Depression Rating Scale (HDRS; 21-item) scores in the non-depressed range (less than 8), and with no more than one clinically significant depressive symptom.

Unaffected MDD Relative Sample:

40 healthy relatives of MDD probands (ages 18-45) will be recruited. Subjects will be screened to ensure that they have no history of psychiatric illness.

Unaffected BD Relative Sample:

Healthy relatives of BD probands (ages 18-45) will be recruited. Subjects will be screened to ensure that they have no history of psychiatric illness.

Healthy Control Samples:

-Healthy subjects (ages 18-45) without a known personal or first-degree family history of psychiatric disorders in first-degree relatives will be selected.

EXCLUSION CRITERIA:

* Any subject who appears incapable of providing informed consent will be excluded from the study.
* Subjects who take effective antidepressant medication
* Subjects must not have taken antidepressant or other medications likely to alter monoamine neurochemistry or cerebrovascular and cardiovascular function for at least 3 months prior to the studies.
* Subjects who have:

  1. psychosis to the extent that the ability to provide informed consent is in doubt
  2. medical or neurological illnesses likely to affect physiology or anatomy, i.e. hypertension, cardiovascular disorders
  3. a history of drug (including benzodiazepines [BZD]) or alcohol abuse within 1 year or a lifetime history of alcohol or drug dependence (DSM IV criteria) longer than 2 years
  4. current pregnancy (as documented by pregnancy testing at screening or at days of the challenge studies)
  5. current breast feeding
  6. smokers
  7. serious suicidal ideation or behavior
  8. general MRI exclusion criteria (e.g., subjects with metallic implants that are ferromagnetic will be excluded from the fMRI scanning). Subjects must exhibit no or only moderate alcohol use. Subjects with current excessive use of alcohol (greater than 4 ounces/day for men and greater than 3 ounces/day for women) are ineligible for participation, as such drug use confounds the results
  9. smokers are ineligible because of the evidence for interactions between nicotine and depression, and the possibility of withdrawal symptoms that may affect behavioral and neural responses to CD
  10. history of suicidality and other axis I diagnoses beside major depressive disorder
  11. lactose intolerance
  12. women not using a reliable contraception method. Finally subjects who have had an upper respiratory tract infection in the last week will be excluded as this may impact sense of smell.
* Subjects beyond age 45
* Individuals whose first major depressive episodes arose after other medical or psychiatric conditions
* Subjects showing significant side effects during AMPT depletion such as dystonic reactions will receive adequate treatment and will be excluded from the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2004-04-19; Study Completion 2011-11-18

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Verhoeff NP, Christensen BK, Hussey D, Lee M, Papatheodorou G, Kopala L, Rui Q, Zipursky RB, Kapur S. Effects of catecholamine depletion on D2 receptor binding, mood, and attentiveness in humans: a replication study. Pharmacol Biochem Behav. 2003 Jan;74(2):425-32. doi: 10.1016/s0091-3057(02)01028-6. PMID 12479964
- [Background] Verhoeff NP, Kapur S, Hussey D, Lee M, Christensen B, C Psych, Papatheodorou G, Zipursky RB. A simple method to measure baseline occupancy of neostriatal dopamine D2 receptors by dopamine in vivo in healthy subjects. Neuropsychopharmacology. 2001 Aug;25(2):213-23. doi: 10.1016/S0893-133X(01)00231-7. PMID 11425505
- [Background] Lambert G, Johansson M, Agren H, Friberg P. Reduced brain norepinephrine and dopamine release in treatment-refractory depressive illness: evidence in support of the catecholamine hypothesis of mood disorders. Arch Gen Psychiatry. 2000 Aug;57(8):787-93. doi: 10.1001/archpsyc.57.8.787. PMID 10920468